CLINICAL TRIAL: NCT03872141
Title: Objective Evaluation of Paclitaxel/Docetaxel-induced Neuropathy in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000020709
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Chemotherapy Induced Peripheral Neuropathy; Paclitaxel Induced Neuropathy
Keywords: neuropathy; taxane; docetaxel
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with stage I-III breast cancer: Patients with Stage I-III breast cancer who will receive paclitaxel or docetaxel treatments as part of their standard of care adjuvant or neoadjuvant therapy are eligible for this study.
  Interventions: Diagnostic Test: Quantitative measures of reduction in Chemotherapy Induced Neuropathy (CIPN) and Cognitive Impairment (CICI) in patients with stage I-III breast cancer

INTERVENTIONS:
Diagnostic Test: Quantitative measures of reduction in Chemotherapy Induced Neuropathy (CIPN) and Cognitive Impairment (CICI) in patients with stage I-III breast cancer — Quantitative measures that include additional aspects of peripheral neuropathy, such as pain, thermal allodynia, numbness and tingling are needed. We propose to evaluate several pharmacodynamics biomarkers in patients before and during chemotherapy: changes in nerve conduction velocity and amplitude, quantitative sensory testing (QST), computer based cognitive assessment, and rate of drop-out from treatment. The tests from this list that best correlate with decreased CIPN would be added to EORTC QLQ-CIPN20 scores and will provide an early indication of CIPN and/or CICI.

SUMMARY:
The purpose of this prospective, non-interventional study is to perform neurological and cognitive assessment of breast cancer patients who receive standard of care single agent weekly paclitaxel docetaxel chemotherapy to determine the onset and severity of chemotherapy induced neuropathy (CIPN) and cognitive impairment (CICI).

DETAILED DESCRIPTION:
The purpose of this prospective, non-interventional study is to perform neurological and cognitive assessment of breast cancer patients who receive standard of care single agent weekly paclitaxel or docetaxel chemotherapy to determine the onset and severity of chemotherapy induced neuropathy (CIPN) and cognitive impairment (CICI).

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 to 70 with histologically confirmed clinically stage I-III breast cancer who will receive weekly paclitaxel (80 mg/m2) or docetaxel (60-100mg/m2) chemotherapy as part of their routine care.

Exclusion Criteria:

* diabetes mellitus
* prior history of neuropathy or symptoms of numbness or peripheral pain, or prior neurotoxic chemotherapy.
* current symptoms of numbness and neuropathic pain
* treatment for bipolar disease
* treatment or concomitant use of common medications used to treat neuropathic pain, such as amitriptyline, gabapentin, pregabalin, duloxetine, for any indication
* limited English that would preclude understanding and completion of the study questionnaires
* pregnancy
* life expectancy <12 weeks
* participation in other research studies either concurrent with or within 30 days prior to participation in this study may be an exclusion criteria

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — women with histologically confirmed clinically stage I-III breast cancer
Study Population: Patients with Stage I-III breast cancer who will receive paclitaxel (80 mg/m2) or docetaxel (60-100mg/m2) as part of their standard of care adjuvant or neoadjuvant therapy are eligible for this study. Women of all races and ethnic groups will be eligible for this trial.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Verbal Memory Test | 20 minutes
  The phrase "Shopping List Learning" is displayed on screen. The pre-task on-screen instructions tell the test supervisor to start this task with the screen facing the supervisor so that the subject cannot see the screen. There are 3 initial rounds of this test. In the first round, the subject is told by the test supervisor: "In this task, I am going to read you a shopping list. I would like you to remember as many items from this list as possible.Total number of correct responses made in remembering the 16 word list on three consecutive learning trials. (Higher score = better performance)
Information processing psychomotor function | 20 minutes
  The pre-task on-screen instructions ask: "Has the card turned over?" The test supervisor reads the full instructions to the subject from the test supervisor script. To begin the task, a playing card is presented in the center of the screen. The card will flip over so it is face up. As soon as it does, the subject must press the "Yes" key. The card will go to the back of the pack and the subject must press the "Yes" key as soon as the next card flips over and so on. The subject will practice until they reach the required number of responses, or until the practice period expires. Then, on screen instructions for the real test are presented. The test supervisor or subject must press the "Enter" key to begin the real test.
  Speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score = better performance
Identification | 20 minutes
  To begin the task, the test supervisor or subject must press the "Enter" key. A playing card is presented in the center of the screen. The card will flip over so it is face up. As soon as it does this the subject must decide whether the card is red or not. If it is red they should press "Yes", if it is not red they should press "No". The subject will practice until they reach the required number of responses, or until the practice period expires. Then, on screen instructions for the real test are presented. The subject should be encouraged to work as quickly as they can and be as accurate as they can.
  Low score = better performance.
Visual Working Memory | 20 minutes
  The pre-task on-screen instructions ask: "Is the previous card the same?" The test supervisor will read full instructions to the subject from the test supervisor script. To begin the task,a playing card is presented in the center of the screen. As soon as it does the subject must decide whether or not the card is the same as the previous one. As this is the first card in this task, the first answer is always "No". Each time a card is revealed, the subject must decide whether the card presented is the same as the one immediately presented previously, and respond by pressing the "Yes" or "No" key. The subject should be encouraged to work as quickly as they can and be as accurate as they can.
  Speed of performance; mean of the log10 transformed reaction times for correct responses.
  Lower score = better performance
Visual Learning Memory | 20 minutes
  The pre-task on-screen instructions ask: "Have you seen this card before in this task?" The test supervisor will read full instructions to the subject from the test supervisor script.
  To begin the task, the test supervisor or subject must press the "Enter" key. A playing card is presented in the center of the screen. As soon as it does the subject must decide whether or not the same card has been seen before in this task. Therefore, the first answer is always "No". Each time a card is revealed, the subject must decide whether they have been shown that card before in this task and respond by pressing the "Yes" or "No" key. The subject should be encouraged to work as quickly as they can and be as accurate as they can.
  Accuracy of performance; arcsine transformation of the proportion of correct responses.
  Higher score = better performance
Verbal Memory Test - Delay | 20 minutes
  The test supervisor presses the "ENTER" key to begin and instructs the subject "Tell me as many of the items on the shopping list that you learned earlier as you can remember now." They then note all of the items recalled by the subject by clicking/touching the corresponding button on screen with the stylus or mouse.
  Total number of correct responses made in recalling the 16 words learned previously after a delay. (Higher score = better performance

SECONDARY OUTCOMES:
To correlate neuronal calcium sensor 1 (NCS1) levels with development of chemotherapy-induced peripheral neuropathy (CIPN) and/or chemotherapy-induced cognitive impairment (CICI) in human patients. | baseline
  Blood samples will be collected in heparinized tubes before the first paclitaxel/docetaxel treatment (baseline). We will collect approximately 20 mL of blood from each subject. White blood cells will be isolated using standard procedures. NCS1 levels will be assessed by Western blot analysis and by qPCR. Additional parameters will be monitored, especially if the variability in NCS1 levels is large. Parameters will be chosen from our understanding of the biochemical pathways identified in the Ehrlich laboratory as part of a separate on-going basic project. The prospective NCS1 values will be correlated with the assessment of CIPN and CICI in each patient obtained in Aim 1.
To correlate NCS1 levels with development of CIPN and/or CICI in human patients. | 6 weeks
  Blood samples will be collected in heparinized tubes before the first paclitaxel/docetaxel treatment and at week 6 during therapy. We will collect approximately 20 mL of blood from each subject. White blood cells will be isolated using standard procedures. NCS1 levels will be assessed by Western blot analysis and by qPCR. Additional parameters will be monitored, especially if the variability in NCS1 levels is large. Parameters will be chosen from our understanding of the biochemical pathways identified in the Ehrlich laboratory as part of a separate on-going basic project. The prospective NCS1 values will be correlated with the assessment of CIPN and CICI in each patient obtained in Aim 1.
To correlate NCS1 levels with development of CIPN and/or CICI in human patients. | 12 weeks
  Blood samples will be collected in heparinized tubes before the first paclitaxel/docetaxel treatment at week 12 during therapy. We will collect approximately 20 mL of blood from each subject. White blood cells will be isolated using standard procedures. NCS1 levels will be assessed by Western blot analysis and by qPCR. Additional parameters will be monitored, especially if the variability in NCS1 levels is large. Parameters will be chosen from our understanding of the biochemical pathways identified in the Ehrlich laboratory as part of a separate on-going basic project. The prospective NCS1 values will be correlated with the assessment of CIPN and CICI in each patient obtained in Aim 1.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ehrlich, PhD, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Center, New Haven, Connecticut, United States